CLINICAL TRIAL: NCT03553095
Title: Comparing Inflammatory Markers in Patients With and Without Depression With Chronic Periodontitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Maninder Kaur, Principal Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-300000426; UAB-Perio (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Chronic Periodontitis; Depression
MeSH Terms: conditions — Chronic Periodontitis; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chronic Periodontitis and Depression Medications (Active Comparator): Patients with clinically diagnosed depression taking (SSRIs, NDRIs, SNRIs, tricyclic antidepressants) and with chronic periodontitis
  Interventions: Procedure: Periodontal Surgery
- Chronic Periodontitis without Depression Medications (Active Comparator): Patients with clinically diagnosed depression not taking any antidepressants (SSRIs NDRIs, SNRIs and Tricyclic antidepressants) and with chronic periodontitis
  Interventions: Procedure: Periodontal Surgery
- Chronic Periodontitis (Active Comparator): Patients without depression, not taking any antidepressants and with chronic periodontitis
  Interventions: Procedure: Periodontal Surgery

INTERVENTIONS:
Procedure: Periodontal Surgery — Samples will be collected from patient in need of periodontal therapy (surgical procedures i.e. gum surgery, tooth extraction and or dental implant surgery). As standard during this procedures remnant tissue is otherwise discarded.

SUMMARY:
This study will evaluate whether use of antidepressants can reduce gingival inflammation in patients with periodontal (gum) disease.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate whether use of antidepressants can reduce gingival inflammation in patients with periodontal (gum) disease. This study will also investigate the link between oral and systemic inflammation in patients diagnosed with depression and periodontal disease. Researcher will collect gingival crevicular fluid, plaque, tissue and blood serum samples to evaluate the link between these two diseases. The collection of gingival crevicular fluid, plaque and blood serum is relatively non-invasive, elicits minimal discomfort and does not require use of any anesthesia. The soft tissue sample will be collected as part of an otherwise planned periodontal surgical procedure under local anesthesia. In periodontal therapy (surgical procedures i.e. gum surgery, tooth extraction and or dental implant surgery) there is enough availability of remnant tissue for the collection of samples, which is otherwise discarded.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Must be a patient of the UAB Dental School
* Able to read and understand informed consent document
* Good general health as evidenced by medical history
* Minimum of 18 teeth, excluding third molars
* Having moderate to severe periodontal disease according to AAP definition (teeth ≥5 mm PD and ≥3 mm CAL)
* Having >30 percent bleeding sites upon probing
* Patients taking depression medication with chronic periodontitis
* Patients without depression with chronic periodontitis
* Patients who have not had a dental cleaning in the past 3 months prior to procedure
* Patients scheduled for surgical procedures (i.e. gum surgery, tooth extraction, or dental implants)

Exclusion Criteria:

* Non-English speaking
* Less than 18 years old
* Smokers/tobacco users (>10 cigarettes/day)
* Any dental condition that requires immediate treatment, such as emergency care
* Chronic use (≥3 times/week) of anti-inflammatory medications (e.g., non-steroidal anti-inflammatory drugs, steroids). Low-dose aspirin (less than 325 mg daily)
* Immunocompromised subjects
* Any medical history or any concomitant medication that might affect the assessment of the study treatment or periodontal tissues, such as uncontrolled diabetes, nifedipine, phenytoin (Dilantin), subjects with arthritis and morbidly obese (BMI ≥ 40)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Gingival crevicular fluid (GCF) | baseline to 1 week
  Measuring oral inflammatory markers in Gingival crevicular fluid (GCF) in patient with chronic periodontitis.

SECONDARY OUTCOMES:
Plaque | baseline to 1 week
  Analyze the type of bacteria that is present in patient with chronic periodontitis.

OTHER OUTCOMES:
Soft tissue | baseline to 1 week
  Analyze the immune cells in patient with chronic periodontitis.
Blood Serum | baseline to 1 week
  Analyze the systemic inflammatory markers in patient with chronic periodontitis.
Patient Health Questionnaire 8 (PHQ8) | baseline to 1 week
  Measure depression status in patient with chronic periodontitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Unversity of Alabama at Birmingham, School of Dentistry, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No